CLINICAL TRIAL: NCT01053585
Title: Combined Magnetic Resonance Imaging and High Resolution Manometry Studies
Brief Title: Structure and Function of the Gastro-esophageal Junction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Dr. Mark Fox, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EK 1361
Record Dates: First submitted 2009-07-21; First posted 2010-01-21 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastro-esophageal junction, reflux, insertion angle, magnetic resonance imaging, manometry
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen (Active Comparator): Baclofen suspension 40mg (single dose 90 minutes prior to physiologic measurement)
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Placebo suspension (single dose 90 minutes prior to physiologic measurement)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Baclofen suspension 40mg (single dose 90 minutes prior to physiologic measurement)
  Arms: Baclofen
Drug: Placebo — Placebo single 'dose' 90 minutes prior to study
  Arms: Placebo

SUMMARY:
Aims of research project:

To identify key features of the gastro-esophageal junction (structure and function) that protects the esophagus from gastro-esophageal reflux investigated by combined high resolution manometry and magnetic resonance imaging.

Hypothesis:

1. Functional factors including GEJ function (e.g. sphincter pressure) and proximal gastric distension determine whether or not TLESR occurs; however
2. Structural factors including separation of GEJ anatomy, intra-gastric distribution of the meal and secretions determine whether TLESR is accompanied by no reflux event, gas reflux (belching) or reflux of ingested food and gastric secretion ('true reflux').
3. Initial findings by descriptive studies in healthy volunteers (study #1) and patients with mild to moderate gastro-esophageal reflux disease (study #2) will be further interrogated by a randomized, double-blind control trial of baclofen in patients with GORD; a medication that inhibits reflux by effects on GOJ function (study #3) .

ELIGIBILITY:
Inclusion criteria:

Study #1:

* healthy male and female volunteers
* aged at least 18 and not more than 49 y
* no history of gastrointestinal symptoms
* able to communicate well with the investigators and to comply with the requirements for the entire study
* who provided written informed consent before participating in the study, after being given a full description of the trail.

Study #2 and #3:

* male and female patients with mild to moderate gastro-oesophageal reflux disease defined by presence of (1) reflux symptoms (2) pathological esophageal acid exposure between 5-10% on 24 hour ambulatory testing
* aged at least 18 and not more than 49 y
* no history of gastrointestinal symptoms
* able to communicate well with the investigators and to comply with the requirements for the entire study
* who provided written informed consent before participating in the study, after being given a full description of the trail.

Exclusion criteria:

* with present psychiatric disorders or mental impairment limiting the ability to comply with study requirements
* with use of medications influencing upper GI motility within one week of the study (i.e. beta- blocker, calcium channel blockers, nitrates, prokinetic drugs, macrolide antibiotics)
* with regular intake of medication; occasional use of analgesic e.g. aspirin, paracetamol is allowed
* with symptoms or a history of gastrointestinal disease other than gastro-esophageal reflux disease (in study #2 and #3)
* suffering from known liver, kidney, cardiovascular, neurological or pulmonary disease
* with any evidence of infectious disease
* with evidence or history of drug or alcohol abuse
* with insufficient knowledge of the German language • who, for any reason, are unable to complete the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Gastro-oesophageal insertion angle, contact span (of stomach on oesophagus) | Pre- and post-meal ingestion
  Gastro-oesophageal morphology from MRI imaging: insertion angle, contact span (of stomach on oesophagus) assessed from 3D models of stomach reconstructed from MRI imaging

SECONDARY OUTCOMES:
gastric emptying | post-meal
  dynamic change in gastric and meal volumes over course of study assessed from MRI imaging. gastric emptying assessed from complete data set
gastric accommodation | post-meal
  dynamic change in gastric and meal volumes over course of study assessed from MRI imaging. gastric accommodation assessed from complete data set
number of reflux events | post-meal
  assessed by presence of common cavity events on (high resolution) manometry

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Division of Gastroenterology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Curcic J, Roy S, Schwizer A, Kaufman E, Forras-Kaufman Z, Menne D, Hebbard GS, Treier R, Boesiger P, Steingoetter A, Fried M, Schwizer W, Pal A, Fox M. Abnormal structure and function of the esophagogastric junction and proximal stomach in gastroesophageal reflux disease. Am J Gastroenterol. 2014 May;109(5):658-67. doi: 10.1038/ajg.2014.25. Epub 2014 Mar 4. PMID 24589669